CLINICAL TRIAL: NCT06654024
Title: Assessment of Urinary Congophilia As an Indicator of Disease Activity of Lupus Nephritis
Brief Title: Urinary Congophilia As an Indicator of Activity of Lupus Nephritis
Acronym: lupus nephriti
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Setohy Hussein Ali, assistant lecturer, Assiut University
Other Study IDs: urinary congophilia in LN
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Lupus Nephritis (LN)
Keywords: congophilia; lupus nephritis; congo red
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Evaluation of the impact of SLE on urinary levels of congophilia and their relationship to renal histopathology and activity of lupus nephritis (LN)

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is an inflammatory autoimmune disease that can affect all body organs. The reported lifetime incidence of lupus nephritis (LN) in SLE patients is 20%- 60% and it is histologically evident in most SLE patients, even without clinical manifestations of kidney disease .

Lupus nephritis is associated with higher mortality , as within 5 years of diagnosis, between 10 and 30 percent of these people develop end-stage renal disease . Early detection and treatment of lupus nephritis can significantly improve renal outcomes and decrease overall mortality .

Endoplasmic reticulum (ER) stress proteins, which act as protein quality control factors in the secretory pathway in the cell are induced by ER stress in inflammatory lesions, and also participate in autoimmunity and inflammation processes, ER stress proteins are expressed not only in the ER but also occasionally at the cell surface that plays pathophysiological roles in autoimmune and inflammatory diseases as pro- or anti-inflammatory factors, Protein folding is easily impaired (misfolding) by different cytotoxic stresses as inflammation or hypoxia , that may contribute to disease pathogenesis by either reducing the biological activity of the protein or due to toxicity by the misfolded proteins, The detection of the abnormally misfolded proteins using the Congo red stain is referred to as congophilia, Urinary congophilia was assessed by Congo Red Dot Blot (CRDB) Assay Congo red is a synthetic diazo dye with specific affinity for β-sheets of amyloid fibrils of misfolded proteins, In addition to the simplicity of congophilia based dot blot technique, the non-invasiveness of the method is useful in adapting the CRDB assay for self-collected urine samples.

One previous study in pregnant females with lupus nephritis said that urinary congophilia has a diagnostic value in patients with lupus nephritis and can be used as a reliable marker of disease activity as the presence of urinary congophilia biomarker is related to disease activity rather than pregnancy.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients ≥ 18 years old that were diagnosed with SLE according to EULAR/ACR classification criteria 2019 for SLE, and lupus nephritis based on renal biopsy or active urinary sediment (proteinuria or hematuria )

Exclusion Criteria:

* Any patient has evidence of nephritis that may cause proteinuria as diabetes mellitus and any other causes of glomerulonephritis other than lupus nephritis
* pregnant females with lupus nephritis and hypertensive disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients ≥ 18 years old that were diagnosed with SLE according to EULAR/ACR classification criteria 2019 for SLE, and lupus nephritis based on renal biopsy or active urinary sediment (proteinuria or hematuria ) ,all are included in this study
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
urinary congophilia level in patient with lupus nephritis is a marker for disease activity | baseline
  Urinary congophilia levels increase in patients with lupus nephritis so that it can be used as a non-invasive urinary marker of lupus nephritis activity.

CONTACTS AND LOCATIONS:
Overall Officials: Radwa Awad Abdelhafiz, PhD doctorate, Study Director — assuit university, faculty of medicine; Samir Kamal Abd elhameed, Professor, Study Director — assuit university, faculty of medicine
Locations (1):
- Assuit University ,Faculty of Medicine, Assute, Assute, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prasanwong T, Laoharojvongsa N, Pongpanich K, Satirapoj B, Charoenpitakchai M. Pathological assessment of activity and chronicity indices in lupus nephritis patients. Asian Arch Path. 2020;2:3-13.
- [Background] Aringer M. EULAR/ACR classification criteria for SLE. Semin Arthritis Rheum. 2019 Dec;49(3S):S14-S17. doi: 10.1016/j.semarthrit.2019.09.009. PMID 31779843
- [Background] Younis D, Shemies RS, El-Kannishy G, Mosbah A, Zakaria M, Awadalla A, et al. # 5383 THE PREDICTIVE VALUE OF URINARY CONGOPHILIA AS A BIOMARKER IN PREGNANT AND NON-PREGNANT WOMEN WITH LUPUS NEPHRITIS. Nephrology Dialysis Transplantation.
- [Background] Khaliq OP, Phoswa WN, Moodley J. The effectiveness of the Congo Red Dot paper test in hypertensive disorders of pregnancy: A systematic review and meta-analysis. Front Reprod Health. 2023 Feb 13;5:1120937. doi: 10.3389/frph.2023.1120937. eCollection 2023. PMID 36864848
- [Background] Buhimschi IA, Nayeri UA, Zhao G, Shook LL, Pensalfini A, Funai EF, Bernstein IM, Glabe CG, Buhimschi CS. Protein misfolding, congophilia, oligomerization, and defective amyloid processing in preeclampsia. Sci Transl Med. 2014 Jul 16;6(245):245ra92. doi: 10.1126/scitranslmed.3008808. PMID 25031267
- [Background] Nagarajappa C, Rangappa SS, Suryanarayana R, Balakrishna S. Urinary congophilia in preeclampsia: Experience from a rural tertiary-care hospital in India. Pregnancy Hypertens. 2018 Jul;13:83-86. doi: 10.1016/j.preghy.2018.05.006. Epub 2018 May 14. PMID 30177078
- [Background] Morito D, Nagata K. ER Stress Proteins in Autoimmune and Inflammatory Diseases. Front Immunol. 2012 Mar 15;3:48. doi: 10.3389/fimmu.2012.00048. eCollection 2012. PMID 22566930
- [Background] Kostopoulou M, Adamichou C, Bertsias G. An Update on the Diagnosis and Management of Lupus Nephritis. Curr Rheumatol Rep. 2020 Jun 4;22(7):30. doi: 10.1007/s11926-020-00906-7. PMID 32500443
- [Background] Mok CC, Teng YKO, Saxena R, Tanaka Y. Treatment of lupus nephritis: consensus, evidence and perspectives. Nat Rev Rheumatol. 2023 Apr;19(4):227-238. doi: 10.1038/s41584-023-00925-5. Epub 2023 Mar 2. PMID 36864291
- [Background] Gasparotto M, Gatto M, Binda V, Doria A, Moroni G. Lupus nephritis: clinical presentations and outcomes in the 21st century. Rheumatology (Oxford). 2020 Dec 5;59(Suppl5):v39-v51. doi: 10.1093/rheumatology/keaa381. PMID 33280015
- [Background] Zen M, Salmaso L, Barbiellini Amidei C, Fedeli U, Bellio S, Iaccarino L, Doria A, Saia M. Mortality and causes of death in systemic lupus erythematosus over the last decade: Data from a large population-based study. Eur J Intern Med. 2023 Jun;112:45-51. doi: 10.1016/j.ejim.2023.02.004. Epub 2023 Feb 9. PMID 36774306
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Lupus Nephritis Work Group. KDIGO 2024 Clinical Practice Guideline for the management of LUPUS NEPHRITIS. Kidney Int. 2024 Jan;105(1S):S1-S69. doi: 10.1016/j.kint.2023.09.002. No abstract available. PMID 38182286